CLINICAL TRIAL: NCT04642209
Title: Platelet Aggregometry to Drive the Surgical Timing in Elderlies With Hip Fracture and Receiving Clopidogrel.
Brief Title: Aggregometry in Elderlies With Hip Fracture and Receiving Clopidogrel
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Federico Longhini, Director, University Magna Graecia
Other Study IDs: Teg-Femur
Record Dates: First submitted 2020-11-12; First posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Hip Fractures; Clopidogrel, Poor Metabolism of; Anesthesia
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aggregometry: surgical timing will be guided by the results obtained by aggregometry
  Interventions: Device: Aggregometry

INTERVENTIONS:
Device: Aggregometry — After evaluation at the Emergency Department the anesthesiologist immediately collects a sample of blood for TEG with ADP Platelet Mapping test.
  If both MA-ADP and platelets aggregation (%) are within normal values (i.e. ≥45 mm and ≥83%, respectively), the patient could be considered as candidate for immediate surgery (within 48 hours) with neuraxial anesthesia.
  If MA-ADP and/or platelets aggregation (%) are lower than normal values, the Nottingham Hip Fracture Score (NHFS) is computed, to predict the 30-day mortality after hip fracture surgery. If NHFS is ≥4 (high risk), the patient will undergo to general anesthesia and peripheral antalgic block, to perform surgery within 48 hours. In case of low risk for mortality (i.e. a NHFS <4), surgery will be postponed until the normalization of both MA-ADP and platelet aggregation.

SUMMARY:
In elderly patients, hip fracture should be surgically treated within 48 hours from admission, since its deferral worsens the mortality. However, sometimes patients are affected by cardiovascular or cerebral comorbidities, deeming necessary the use of antiplatelets and/or anticoagulant therapies. Clopidogrel is a second-generation thienopyridine antiplatelet drug which exerts its effect by the inhibition of the platelet's purinergic receptor P2Y12 preventing adenosine diphosphate (ADP) from stimulating it. Guidelines recommend to withhold clopidogrel for 5 days before the possibility to perform neuraxial anesthesia, which is frequently the optimal perioperative management of a fragile patient. It should be mentioned however that around 30% of patients are resistant to clopidogrel and they show a normal platelet reactivity despite the antiplatelet therapy. Therefore, in principle, these patients do not require to defer surgery. We have therefore hypothesized that some patients taking clopidogrel might anticipate surgery before 5 days and within 48 hours, following a protocol based on the assessment of coagulation and platelet aggregation through thromboelastography (TEG) in combination with an ADP Platelet Mapping assay kit.

After hospital admission for femur fracture, eligible patients would be evaluated by the anesthesiologist and the orthopedic physicians for anesthesia and surgery. Immediately a sample of blood should be collected for TEG with ADP Platelet Mapping test. If both MA-ADP and platelets aggregation (%) will be within normal values, the patient could be considered as candidate for immediate surgery (within 48 hours) with neuraxial anesthesia and ultrasound-guided antalgic femoral nerve block. If MA-ADP and/or platelets aggregation (%) are lower, risk for mortality should be assessed. If the patient would be considered at high risk for mortality, he/she would undergo to general anesthesia and peripheral antalgic block to not postpone surgery. Otherwise, surgery would be postponed until the normalization of both MA-ADP and platelet aggregation.

DETAILED DESCRIPTION:
Hip fracture is an established and recognized health problem associated with the age of the population. In the elderly, it is essential that surgery for hip fractures would be performed within 48 hours from admission. Whenever delayed beyond 48 hours, the probability of 30-day mortality increases by 41% and the odds of one-year mortality by 32%.

Neuraxial anesthesia and/or peripheral nerve block are generally preferred in elderlies. However, cardiovascular and/or cerebral comorbidities require antiplatelets therapies at home. This treatment precludes the possibility of an optimal anesthesiologic strategy (i.e., loco-regional anesthesia) within the recommended surgical timing. Therefore, an individual approach is required to balance the risk of drugs continuation/cessation on major cardiovascular events and on peri-operative bleeding.

Clopidogrel is a second-generation thienopyridine antiplatelet drug, that exerts its effect by the inhibition of the platelet's purinergic receptor P2Y12, preventing adenosine diphosphate (ADP) from stimulating it. In patients needing surgery, guidelines recommend withholding clopidogrel 5 days before. However, around 30% of patients are resistant to clopidogrel for several reasons. Patients resistant to clopidogrel may be identify through the thromboelastography (TEG). TEG is a resonance-frequency viscoelastic point-of-care diagnostic system that assesses hemostasis and response to antiplatelet therapy, in combination with the ADP Platelet Mapping assay kit.

It has been hypothesized that the assessment of platelet aggregation with TEG and ADP Platelet Mapping may identify patients resistant to clopidogrel, not requiring to wait for 5 days for hip replacement surgery. We have therefore designed this protocol to guide anesthesiologists in the management of elderlies receiving clopidogrel and requiring surgery for hip fracture. The aim of this pilot study is to evaluate if in a small population of patients, our protocol based on platelet function monitoring would anticipate surgery within 48 hours at least in 70% of elderly patients receiving clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* all patients older than 65 years/old
* admission to the hospital for suspected traumatic femur fracture
* home therapy with clopidogrel 75 mg/die at home

Exclusion Criteria:

* pre-existing coagulopathies
* assumption of any anticoagulant oral therapy
* platelet count <100.000 mcL
* pre-existing liver disease
* known autoimmune diseases
* presence of hematological malignancies

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients older than 65 years/old, admitted to the hospital for suspected traumatic femur fracture receiving clopidogrel 75 mg/die at home were consecutively included in the pilot study.
  Patients with one or more of the following criteria were excluded: 1) pre-existing coagulopathies; 2) assumption of any anticoagulant oral therapy; 3) platelet count <100.000 mcL; 4) pre-existing liver disease; 5) known autoimmune diseases; 6) presence of hematological malignancies.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2020-12-15 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Patients undergoing to hip replacement surgery | within 48 hours from hospital admission
  Number of patients undergoing to hip replacement surgery within 48 hours from hospital admission

SECONDARY OUTCOMES:
Occurrence of peri or post-operative complications | 28 days from admission
  Occurrence of peri or post-operative complications, such as postoperative myocardial infarction, thromboembolism, and postoperative confusion
Occurrence of intra-operative hypotension | During surgery
  Reduction of mean arterial pressure by 10% from baseline
Presence of post-operative bleeding | Within 48 hours after surgery
  Presence of post-operative bleeding greater than 600 ml, considered as clinically relevant

CONTACTS AND LOCATIONS:
Overall Officials: Federico Longhini, MD, Study Chair — Magna Graecia University, Anesthesia and Intensive Care Unit
Locations (1):
- Federico Longhini, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: Yes
data will be shared on reasonable request to the corresponding author
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: After study publication

REFERENCES:
- [Background] Bottle A, Aylin P. Mortality associated with delay in operation after hip fracture: observational study. BMJ. 2006 Apr 22;332(7547):947-51. doi: 10.1136/bmj.38790.468519.55. Epub 2006 Mar 22. PMID 16554334
- [Background] Kristensen SD, Knuuti J, Saraste A, Anker S, Botker HE, De Hert S, Ford I, Gonzalez Juanatey JR, Gorenek B, Heyndrickx GR, Hoeft A, Huber K, Iung B, Kjeldsen KP, Longrois D, Luescher TF, Pierard L, Pocock S, Price S, Roffi M, Sirnes PA, Uva MS, Voudris V, Funck-Brentano C; Authors/Task Force Members. 2014 ESC/ESA Guidelines on non-cardiac surgery: cardiovascular assessment and management: The Joint Task Force on non-cardiac surgery: cardiovascular assessment and management of the European Society of Cardiology (ESC) and the European Society of Anaesthesiology (ESA). Eur J Anaesthesiol. 2014 Oct;31(10):517-73. doi: 10.1097/EJA.0000000000000150. No abstract available. PMID 25127426
- [Background] Warlo EMK, Arnesen H, Seljeflot I. A brief review on resistance to P2Y12 receptor antagonism in coronary artery disease. Thromb J. 2019 May 20;17:11. doi: 10.1186/s12959-019-0197-5. eCollection 2019. PMID 31198410
- [Background] Tarrant SM, Kim RG, McGregor KL, Palazzi K, Attia J, Balogh ZJ. Dual Antiplatelet Therapy and Surgical Timing in Geriatric Hip Fracture. J Orthop Trauma. 2020 Oct;34(10):559-565. doi: 10.1097/BOT.0000000000001779. PMID 32304474
- [Background] Yang Z, Ni J, Long Z, Kuang L, Gao Y, Tao S. Is hip fracture surgery safe for patients on antiplatelet drugs and is it necessary to delay surgery? A systematic review and meta-analysis. J Orthop Surg Res. 2020 Mar 12;15(1):105. doi: 10.1186/s13018-020-01624-7. PMID 32164755
- [Background] Price MJ, Walder JS, Baker BA, Heiselman DE, Jakubowski JA, Logan DK, Winters KJ, Li W, Angiolillo DJ. Recovery of platelet function after discontinuation of prasugrel or clopidogrel maintenance dosing in aspirin-treated patients with stable coronary disease: the recovery trial. J Am Coll Cardiol. 2012 Jun 19;59(25):2338-43. doi: 10.1016/j.jacc.2012.02.042. PMID 22698488
- [Derived] Tescione M, Vadala E, Marano G, Battaglia E, Bruni A, Garofalo E, Longhini F, Rovida S, Polimeni N, Squillaci R, Lascala S, Franco G, Labate D, Caracciolo M, Macheda S. Platelet aggregometry for hip fracture surgery in patients treated with clopidogrel: a pilot study. J Clin Monit Comput. 2022 Jun;36(3):823-828. doi: 10.1007/s10877-021-00714-z. Epub 2021 May 6. PMID 33956283